CLINICAL TRIAL: NCT04445480
Title: The Benefit of Popliteal Sciatic Nerve Block for Lower Limb Angioplasty in Critical Limb Ischemia: a Randomised Controlled Trial
Brief Title: Popliteal Block for Lower Limb Angioplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SI198/2019
Record Dates: First submitted 2020-03-04; First posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Angioplasty; Anaesthesia and Analgesia
Keywords: popliteal block; chronic limb ischemia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Popliteal block group (Experimental)
  Interventions: Procedure: Popliteal block
- Control group (Active Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Procedure: Popliteal block — Sciatic nerve block at popliteal fossa would perform before the participant undergoing angioplasty in experimental arm.
  Arms: Popliteal block group
Other: Control — Sciatic nerve at popliteal fossa would be scanned with the ultrasound. The toothpick would be applied to simulate the procedure of nerve block.
  Arms: Control group

SUMMARY:
Endovascular revascularization is an effective procedure in treatment of chronic critical limb ischemia. The less invasive procedure in high risk patients produce the benefit to the patients. However, some of the patients cannot tolerate local anaesthesia. These patients need sedation or even general anaesthesia, which increase unnecessary risk to the patients. This study is conducted to evaluate the benefit of popliteal sciatic nerve block or popliteal block compare to sedation in critical limb patients undergoing angioplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 20 year-old with chronic ischemic limb pain
* Scheduled for peripheral angioplasty under monitor anaesthesia care
* Expected timing of procedure not more than 3 hours

Exclusion Criteria:

* Age less than 21
* Cannot cooperate with the staff
* Having pain in other areas or both legs
* Contraindicate for nerve block
* Allergy to local anesthetic drugs or sedative drugs

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of general anaesthesia | Five hours

SECONDARY OUTCOMES:
Numerical pain rating scale during procedure | Five hours

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology department, Siriraj Hospital, Mahidol University, Bangkok, Thailand